CLINICAL TRIAL: NCT04530851
Title: Compare Outcome of Enhanced Recovery After Cesarean Surgery and Conventional Care in Rajavithi Hospital
Brief Title: Compare Outcome of Enhanced Recovery After Cesarean Surgery and Conventional Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103/2562
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: To Determine Whether ERAS Can Reduce Length of Stay in Pregnant Women After Cesarean Section
Keywords: ERAS; Cesarean section; Length of stay

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional care (No Intervention): This group is conventional care of pregnant women after Cesarean section
- ERAS protocol (Experimental): This protocol for improve outcome of pregnant women after Cesarean section
  Interventions: Procedure: ERAS

INTERVENTIONS:
Procedure: ERAS — * Counseling
  * H2- antagonist and metroclopramide for prevent aspiration
  * Drink clear liquid until 2 hour before surgery
  * First generation cephalosporin in 60 minute before surgery
  * Clorhexidine for skin cleansing and Povidine for vaginal cleansing
  * Regional anesthesia
  * Keep warming
  * Blunt expansion of uterine incision
  * Do not peritoneal suture and subcuticular suture if less than 2 cm
  * Local wound anesthesia.
  * Paracetamol and NSAIDs for for pain control
  * Early remove catheter and ambulation
  * 5-HT3 antagonist for prevent nausea
  Arms: ERAS protocol

SUMMARY:
Research objective to compare outcome(Length of stay, pain score, opioid drug use, Bowel function and complication ) of ERAS protocol and conventional care in pregnant women after elective cesarean section in Rajavithi hospital.

DETAILED DESCRIPTION:
Research design is Randomized control trial. The pregnant women who go to elective cesarean section don't know the allocation. The group of ERAS protocol was separated from Conventional care in patient care unit.

The Pregnant are randomly in two group. In the ERAS group the pregnant receive the the intervention for preoperative care(Counselin, H2- antagonist and metroclopramide for prevent aspiration, Drink clear liquid until 2 hour before surgery), Intraoperative care (first generation cephalosporin in 60 minute before surgery, Clorhexidine for skin cleansing and Povidine for vaginal cleansing, regional anesthesia, keep warming, blunt expansion of uterine incision, do not peritoneal suture and subcuticular suture if less than 2 cm, local wound anesthesia.), post operative care ( Paracetamol and NSAIDs for for pain control, early remove catheter and ambulation, 5-HT3 antagonist for prevent nausea)

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who scheduled for elective Cesarean section at Rajavithi Hospital

Exclusion Criteria:

* Pregnant women who has preeclampsia with severe feature
* Pregnant women who has diabetes mellitus with uncontrolled blood sugar
* Pregnant women who has blood loss > 1,500 ml after surgery
* Pregnant women who has chrioamnionitis.
* Pregnant women who has severe medical disease
* Pregnant women who has BMI >= 40 kg/m2
* Pregnant women who has placenta adherence.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Compare length of stay of pregnant women after Cesarean section between ERAS protocol and conventional care | 1 year
  The primary outcome is length of stay (Day)

SECONDARY OUTCOMES:
Compare pain of pregnant women after Cesarean section between ERAS protocol and conventional care | 1 year
  The outcome is pain score (visual analogue scale )
Compare opioid use of pregnant women after Cesarean section between ERAS protocol and conventional care | 1 year
  The outcome are opioid use (Meperidine, Tramadol, Morphine)
Compare complication of pregnant women after Cesarean section between ERAS protocol and conventional care | 1 year
  The outcome are complication after surgery such as fever, wound infection, wound dehiscence, metritis
Compare bowel function of pregnant women after Cesarean section between ERAS protocol and conventional care | 1 year
  The outcome is time to passing gas after surgery(hour)

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi hospital, Bangkok, Thailand